CLINICAL TRIAL: NCT06706388
Title: An Open-label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for ATN1 Gene Mutation
Brief Title: Personalized Antisense Oligonucleotide Therapy for a Single Participant with ATN1 Gene Mutation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV0657
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Dentatorubral-Pallidoluysian Atrophy
MeSH Terms: conditions — Myoclonic Epilepsies, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-ATN1-002

INTERVENTIONS:
Drug: nL-ATN1-002 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with dentatorubral-pallidoluysian atrophy (DRPLA) due to a heterozygous pathogenic CAG trinucleotide expansion in ATN1

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with DRPLA due to a heterozygous pathogenic CAG trinucleotide expansion in ATN1

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.
* Genetically confirmed Dentatorubral-pallidoluysian atrophy (DRPLA) due to ATN1 mutation

Exclusion Criteria:

* Use of investigational medication within 5 half-lives of the drug at enrolment
* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.

Ages: 17 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Ataxia | Baseline to 24 months
  Change in mobility and ataxia from baseline to 6-, 12-, 18- and 24-months post nL-ATN1-002 administration as measured by the Scale for Assessment and Rating of Ataxia (SARA).
Ataxia | Baseline to 24 months
  Change in mobility and ataxia from baseline to 6-, 12-, 18- and 24-months post nL-ATN1-002 administration as measured by wrist/ankle accelerometers (peak velocity, peak acceleration, movement entropy).
Ataxia | Baseline to 24 months
  Change in mobility and ataxia from baseline to 6-, 12-, 18- and 24-months post nL-ATN1-002 administration as measured by home gait video assessment (reviewed by blinded rater using gait and stance rating criteria from the SARA).

SECONDARY OUTCOMES:
Seizures | Baseline to 24 months
  Change in seizure frequency and length of seizures, as well as seizure medication use, from baseline to 12- and 24-months post nL-ATN1-002 administration as measured by caregiver seizure diary tracking.
Quality of Life | Baseline to 24 months
  Change in quality of life from baseline to 6-, 12-, 18- and 24-months post nL-ATN1-002 administration as measured by the Activities of Daily Living questionnaire (ADL).
Quality of Life | Baseline to 24 months
  Change in quality of life from baseline to 6-, 12-, 18- and 24-months post nL-ATN1-002 administration as measured by the Caregiver Global Impression of Change questionnaire (CGI-C).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline to 24 months
Incidence of Treatment-Emergent abnormalities in physical and neurological exams [Safety and tolerability] | Baseline to 24 months
Incidence of Treatment-Emergent abnormalities in safety labs (CSF, chemistry, hematology, coagulation, and urinalysis) [Safety and tolerability] | Baseline to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States